CLINICAL TRIAL: NCT07330882
Title: Health Behavior Management Program for Patients With Coronary Heart Disease: A Clinical Study
Brief Title: Health Behavior Management Program for Patients With Coronary Heart Disease
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Principal Investigator, Zhou,Tong, Associate Professor, The First Affiliated Hospital of Bengbu Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FirstAHBBMC
Record Dates: First submitted 2025-11-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Coronary Disease
Keywords: Myocardial Ischemia; Cardiac rehabilitation; Quality of life; Frailty
MeSH Terms: conditions — Coronary Disease; Myocardial Ischemia; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention consists of two parts: Health management model: Establish a "hospital-home" full-process health management service chain based on mobile health. Firstly, cardiac specialist nurses conduct a comprehensive assessment of each patient's cardiac rehabilitation status and implement individualized interventions. The specific intervention procedures are: "Assess the patient's current condition and capabilities - Promote the patient's awareness of the current situation - Develop and revise the cardiac rehabilitation plan - Supervise the implementation of the cardiac rehabilitation plan."
  Interventions: Behavioral: Exercise rehabilitation plan and health management model for patients with coronary heart disease and frailty based on mobile health technology
- Control group (Active Comparator): During the patient's hospital stay and after discharge, cardiovascular internal medical staff provide them with routine medical,nursing services and health education. In terms of basic drug treatment, the principles of secondary prevention for coronary heart disease should be followed. Routine nursing care and health education were delivered through verbal instruction and the "317 Nursing Education Platform." They were also advised to maintain a healthy lifestyle and participate in appropriate physical activities.
  Interventions: Behavioral: Exercise rehabilitation plan and health management model for patients with coronary heart disease and frailty based on mobile health technology

INTERVENTIONS:
Behavioral: Exercise rehabilitation plan and health management model for patients with coronary heart disease and frailty based on mobile health technology — The development, application and evaluation of an innovative health management model for patients with coronary heart disease and frailty based on the "cardiac rehabilitation center" framework, exercise rehabilitation, and new technologies such as "mobile health".

SUMMARY:
Coronary artery disease (CAD) is a major chronic condition severely impacting population health in China. Our previous cohort studies revealed a high comorbidity rate between CAD and frailty, suggesting their interrelated equivalence as clinical syndromes with shared risk factors. In recent years, pilot integrated health management initiatives in China have demonstrated promising outcomes, yet evidence remains scarce regarding patients with concurrent CAD and frailty-a critical gap needing urgent resolution to achieve the "Healthy China 2030" strategic goals.

Building on prior research, this project aims to systematically evaluate existing management models for patients with CAD and frailty, develop a tailored health management framework, and implement it in clinical settings through empirical studies. The model will be optimized according to regional and demographic variations, leveraging cardiac rehabilitation centers, exercise-based interventions, and internet-enabled technologies to enhance coordinated care. By improving exercise efficacy, mitigating frailty progression, and enhancing quality of life, this initiative seeks to establish a robust chronic disease management system. The findings will provide evidence for formulating regional health policy and insurance strategies in Anhui Province, ultimately improving standardized management rates for chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Coronary heart disease;
* Proficiency in smartphone use;
* Absence of visual, auditory, cognitive, or motor impairments.

Exclusion Criteria:

* Inability or unwillingness to provide informed consent;
* Physical or cognitive limitations preventing app operation;
* Inability to attend in-person follow-up visits;
* Concurrent severe comorbidities or malignancies, such as severe valvular heart disease, New York Heart Association class IV heart failure, severe aortic regurgitation, cancer, end-stage renal or liver disease;
* Any other condition that could potentially impede exercise participation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
6MWD | 1month,3 months, 6 months
  Measuring the maximum distance within 6 minutes.
The MOS item short from health survey | 1month,3 months, 6 months
  Quality of life was assessed using the 36-Item Short Form Health Survey questionnaire

SECONDARY OUTCOMES:
Frailty | 1month,3 months, 6 months
  The FRAIL Scale
Grip strength | 1month,3 months, 6 months
  Electronic grip device
Gait speed | 1month,3 months, 6 months
  Stopwatch
Physical activity level | 1month,3 months, 6 months
  The short version self-reported International Physical Activity Questionnaire.
Systolic pressure/Diastolic pressure | 1month,3 months, 6 months
  Calibrated electronic blood pressure monitor
Major cardiovascular adverse events | 1month,3 months, 6 months
  Major Adverse Cardiovascular Events (MACE) were defined as at least one of the following: heart failure, malignant arrhythmia, recurrent angina, recurrent myocardial infarction, cardiogenic shock, cardiac arrest, or sudden cardiac death.
Changes in Blood Lipid Biomarkers | 1 month, 3 months, 6 months
  Changes in blood lipid biomarkers, including triglycerides (TG), total cholesterol (TC), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C), were assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Tong Zhou, Principal Investigator — The First Affiliated Hospital of Bengbu Medical University
Locations (1):
- The First Affiliated Hospital of Bengbu Medical University, Bengbu, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT07330882/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT07330882/ICF_001.pdf